CLINICAL TRIAL: NCT01465399
Title: Randomized Clinical Trial, Controlled With Conventional Treatment, of Efficacy and Safety of Plasma Rich in Growth Factors (PRGF-Endoret) in the Regeneration of Post-extraction Sockets in Simple Extractions of Molars in the Mandible
Brief Title: Plasma Rich in Growth Factors (PRGF-Endoret) in the Regeneration of Post-Extraction Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Eduardo Anitua (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: FIBEA-01-EC/11/ALV; 2019-001167-75 (EudraCT Number)
Record Dates: First submitted 2011-10-27; First posted 2011-11-04 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Post-Extraction Sockets Healing

ARMS (2):
- PRGF-Endoret (Experimental)
  Interventions: Biological: Plasma Rich in Growth Factors PRGF-Endoret
- Conventional treatment (Active Comparator)
  Interventions: Procedure: Conventional closure of the lesion

INTERVENTIONS:
Biological: Plasma Rich in Growth Factors PRGF-Endoret
  Arms: PRGF-Endoret
Procedure: Conventional closure of the lesion
  Arms: Conventional treatment

SUMMARY:
Immediately following tooth removal, a healing process begins that affects the eventual alveolar bone volume and architecture of the alveolar ridge. Satisfactory and timely healing are essential to obtain ideal functional reconstruction. Traumatic removal of a tooth, or a poor healing response, may lead to excessive bone loss delaying tooth replacement, requiring expensive and time-consuming reconstructive surgeries, or even the inability to be corrected. The Plasma Rich in Growth Factors (PRGF-Endoret) has shown its therapeutic potential effect to minimize the consequences of this aggression, promoting the regeneration of both hard and soft involved tissues.

ELIGIBILITY:
Inclusion Criteria:

* subjects of both genders and ≥ 18 years old
* Indication of a simple one molar extraction in the mandible.
* Possibility of observation during the follow-up period.

Exclusion Criteria:

* Unerupted third molars or with horizontal inclination.
* Severe swelling prior to surgery in the areas designated for extraction.
* Suffering an alteration or a serious hematologic disease.
* Be currently undergoing or have received radiotherapy, chemotherapy or immunosuppressive therapy, corticosteroids and/or anticoagulants 30 days prior to inclusion
* In regular treatment with NSAIDs or other anti-inflammatory drugs.
* History of chronic hepatitis or cirrhosis.
* Diabetes mellitus with poor metabolic control (glycosylated hemoglobin >9%)
* Patients undergoing dialysis.
* Presence of malignant tumors, hemangiomas or angiomas in the extraction area.
* History of ischemic heart disease in the last year.
* Pregnancy or planned pregnancy during the study follow-up period.
* Metabolic Bone Disease.
* Patients taking bisphosphonates both orally and intravenously.
* In general, any inability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of regenerated post-extraction sockets | 10-12 weeks

SECONDARY OUTCOMES:
Regenerated bone volume | 10-12 weeks
  Measurement of the regenerated bone volume at final follow-up in relation to the initial post-extraction socket total volume measured by CT-Scanner and expressed as a percentage.
Post-operative pain (VAS) | 3, 7 and 15 days post-extraction
Soft Tissue Healing Index | 3, 7 and 15 days post-extraction
Inflammation | 3, 7 and 15 days post-extraction
  Using a specific 0 to 3 Inflammation Score
Adverse events or complications | 10-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Anitua, MD, DDS, PhD, Study Director — Clinica Dental Eduardo Anitua
Locations (1):
- Clínica Dental Eduardo Anitua, Vitoria-Gasteiz, Spain